CLINICAL TRIAL: NCT06483308
Title: Shortened High-dose Palliative Radiotherapy for Lung Cancer (SHiP-Rt) Study
Brief Title: Shortened High-dose Palliative Radiotherapy for Lung Cancer
Acronym: SHiP-Rt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS631323
Record Dates: First submitted 2024-06-17; First posted 2024-07-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-03

CONDITIONS: Stage IV Lung Cancer
Keywords: Radiotherapy; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy (Other)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy using 30Gy in 6 fractions (alternate days) over 12 days.

SUMMARY:
The SHiP-Rt Study aims to investigate the safety and efficacy of reducing the number of RT fractions and RT duration, compared to the current standard of care (36Gy in 12 fractions over 16 days), by using shortened hypofractionated accelerated palliative radiotherapy (30Gy in 6 alternate-day fractions), aided by contemporary RT planning, verification, and delivery techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patient has locally advanced (stage IIIB or IIIC) or metastatic (stage IV) NSCLC
* Patient is treatment naïve or had limited progression after first-line systemic therapy (using chemotherapy, immunotherapy, or targeted therapy)
* Patient is suitable for high dose palliative RT (36Gy in 12# or 39Gy in 13#)
* Obtained written informed consent for the SHiP-Rt study.
* Patients receiving RT after first-line systemic therapy must have a wash-out period of at least 3 weeks (i.e., 3-4 weeks).
* Treatment naïve patients should be able to proceed to definitive systemic therapy without undue delay, i.e., within 3-4 weeks.

Exclusion Criteria:

* Contraindication for thoracic RT
* Requiring lung RT after second-line systemic therapy for NSCLC
* Has more than 1 cancer that is requiring active treatment
* On cytotoxic treatment for rheumatoid arthritis or connective tissue disorders
* Poor life expectancy, likely less than 6 months
* Patients with difficulty regarding compliance to the study treatment or follow-up
* Previous radiotherapy to the same area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Successful completion of treatment without reporting grade 3-4 oesophagitis, within 4 weeks of completing RT, using CTCAE v4.03. | 4 weeks of completing RT

SECONDARY OUTCOMES:
Toxicity if proposd hypofractionated high dose palliative RT using CTCAE v4.03 | 12 months
Patient reported outcome measures (PROMS) using Quality-of Life Questionnaires (QLQ-C30 & QLQ-LC13) | 12 months
Disease response and progression | 12 months
Cost-savings calculations to compare the proposed treatment regime to the standard of care. | 12 months
Number of participants offered to participate in the study vs how many consent vs how many complete treatment | 12 months
Time to start systemic therapy from recruitment. | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire
  - University Hospitals Coventry and Warwickshire, Coventry, Warwickshire
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - The Shrewsbury and Telford Hospital NHS Trust, Shrewsbury, West Midlands

REFERENCES:
- [Derived] Shrimali RK, Griffin E, Sturgess V, Jones M, Hiller L, Rogers J, Hamilton J, Peebles C, Jones B, Dunn J. Shortened High-dose Palliative Radiotherapy for Lung Cancer (SHiP-Rt): protocol for a single-arm, multicentre, phase II study. BMJ Open. 2026 Feb 2;16(2):e111350. doi: 10.1136/bmjopen-2025-111350. PMID 41628919